CLINICAL TRIAL: NCT04656652
Title: Phase 3 Randomized Study of DS-1062a Versus Docetaxel in Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer (TROPION-LUNG01)
Brief Title: Study of DS-1062a Versus Docetaxel in Previously Treated Advanced or Metastatic Non-small Cell Lung Cancer With or Without Actionable Genomic Alterations (TROPION-LUNG01)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-U301; 2020-004643-80 (EudraCT Number); 2023-509865-19-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-19; First posted 2020-12-07 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Metastatic Non-small Cell Lung Cancer; Advanced Non-small Cell Lung Cancer; Non-small Cell Lung Cancer; DS-1062; Docetaxel; Datopotamab Deruxtecan (Dato-DXd)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-1062a 6.0 mg/kg (Experimental): Participants will be randomized to receive 6.0 mg/kg of DS-1062a.
  Interventions: Drug: DS-1062a
- Docetaxel 75 mg/m^2 (Active Comparator): Participants will be randomized to receive 75 mg/m^2 docetaxel.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: DS-1062a — DS-1062a will be administered as an intravenous (IV) infusion on Day 1 of each 3-week cycle
  Other Names: Datopotamab deruxtecan (Dato-DXd)
  Arms: DS-1062a 6.0 mg/kg
Drug: Docetaxel — Docetaxel will be administered as an IV infusion on Day 1 of each 3-week cycle.
  Arms: Docetaxel 75 mg/m^2

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of DS-1062a versus docetaxel in participants with previously treated advanced or metastatic non-small cell lung cancer (NSCLC) with or without actionable genomic alterations.

DETAILED DESCRIPTION:
This study will evaluate DS-1062a 6.0 mg/kg vs docetaxel 75 mg/m^2 in participants with advanced or metastatic NSCLC with or without actionable genomic alterations (AGAs). Participants without actionable genomic alterations must have been previously treated with platinum-based chemotherapy and α (anti)-programmed cell death 1 (PD-1)/α-programmed cell death ligand 1 (PD-L1) monoclonal antibody, either in combination or sequentially. Participants with AGA must have progressed on or after 1 platinum-containing therapy and 1 to 2 prior lines of approved targeted therapy for the applicable genomic alteration. The study will be divided into 3 periods: Screening Period, Treatment Period, and Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in the study must meet all inclusion criteria within 28 days of randomization into the study.

* Sign and date the inform consent form (ICF) prior to the start of any study specific qualification procedures.
* Adults ≥18 years (if the legal age of consent is >18 years old, then follow local regulatory requirements)
* Life expectancy ≥3 months
* Has pathologically documented Stage IIIB, IIIC, or stage IV NSCLC disease with or without actionable genomic alterations (AGA) at the time of randomization (based on the American Joint Committee on Cancer, Eighth Edition) and meets following criteria for NSCLC:
* Participants without AGA:

  1. Must have documented negative test results for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK).
  2. Must have no known genomic alterations in ROS proto-oncogene 1 (ROS1), neurotrophic tyrosine receptor kinase (NTRK), proto oncogene B-raf (BRAF), mesenchymal-epithelial transition (MET) exon 14 skipping, or rearranged during transfection (RET).
* Participants with AGA must have one or more documented actionable genomic alteration(s): EGFR, ALK, ROS1, NTRK, BRAF, MET exon 14 skipping, or RET.
* Has documentation of radiographic disease progression while on or after receiving the most recent treatment regimen for advanced or metastatic NSCLC.
* Participant without AGA must meet 1 of the following prior therapy requirements for advanced or metastatic NSCLC:

  1. Received platinum-based chemotherapy in combination with α-PD-1/α-PD-L1 monoclonal antibody as the only prior line of therapy.

     * Includes participants who received prior platinum-based/chemotherapy with or without radiotherapy with maintenance α-PD-1/α-PD-L1 monoclonal antibody for Stage III disease and relapsed/progressed within 6 months from the last dose of platinum-based chemotherapy.
     * Includes participants who received prior platinum-based/chemotherapy with or without radiotherapy (with or without maintenance α-PD-1/α-PD-L1 monoclonal antibody) for Stage III disease and subsequently received α-PD-1/α-PD-L1 monoclonal antibody therapy (with or without platinum-based chemotherapy) for recurrent disease.
  2. Received platinum-based chemotherapy and α-PD-1/α-PD-L1 monoclonal antibody (in either order) sequentially as the only 2 prior lines of therapy.
* Participants with AGA must meet the following for advanced or metastatic NSCLC:

  1. Participants who have been treated with 1 or 2 prior lines of applicable targeted therapy that is locally approved for the participant's genomic alteration at the time of screening;

     * Participants who have tumors with EGFR L858R or exon 19 deletion mutations must have received prior Osimertinib.
     * Those who received a targeted agent as adjuvant therapy for early-stage disease must have relapsed or progressed while on the treatment or within 6 months of the last dose OR received at least one additional course of targeted therapy for the same genomic alteration (which may or may not be same agent used in the adjuvant setting) for relapsed/progressive disease.
     * Participants who have been treated with a prior tyrosine kinase inhibitor (TKI ) must receive additional approved targeted therapy, if locally available and clinically appropriate, for the applicable genomic alteration, or the participant will not be allowed in the study.
  2. Participants who have received platinum-based chemotherapy as the only prior line of cytotoxic therapy:

     * One platinum-containing regimen for advanced disease
     * Those who received a platinum-containing regimen as adjuvant therapy for early-stage disease must have relapsed or progressed while on the treatment or within 6 months of the last dose OR received at least one additional course of platinum-containing therapy (which may or may not be same as in the adjuvant setting) for relapsed/progressive disease.
  3. May have received up to one α-PD-1/α-PD-L1 monoclonal antibody alone or in combination with a cytotoxic agent.
* Must undergo a pre-treatment tumor biopsy procedure or if available, tumor tissue previously retrieved from a biopsy procedure performed within 2 years prior to the participant signing informed consent and that has a minimum of 10 × 4 micron sections or a tissue block equivalent of 10 × 4 micron sections may be substituted for the pre-treatment biopsy procedure during Screening. If a documented law or regulation prohibits (or does not approve) sample collection, then such samples will not be collected/submitted
* Measurable disease based on local imaging assessment using RECIST v1.1
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at Screening
* Within 7 days before randomization, has adequate bone marrow, hepatic, and renal function
* Left ventricular ejection fraction (LVEF) ≥50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before randomization
* Adequate blood clotting function defined as international normalized ratio/prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤1.5 × upper limit of normal (ULN)
* Adequate treatment washout period before randomization
* Females of childbearing potential must have a negative serum pregnancy test at screening and must be willing to use highly effective birth control from the time of enrollment up to 7 months after the last dose of DS-1062a or for at least 6 months after the last dose of docetaxel
* Males must be surgically sterile or must use a condom in addition to highly effective birth control if his partners are of reproductive potential from the time of enrollment and for at least 4 months after last dose of DS-1062a or for at least 6 months after the last dose of docetaxel
* Male participants must not freeze or donate sperm from the time of Screening and throughout the study period and for at least 4 months after the last dose of DS-1062a or for at least 6 months after the last dose of docetaxel
* Female participants must not donate, or retrieve for their own use, ova from the time of Screening and throughout the study period and for at least 7 months after the last dose of DS-1062a and for at least 6 months after the last dose of docetaxel

Exclusion Criteria:

* Mixed small-cell lung cancer (SCLC) and NSCLC histology
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study. Participants with treated brain metastases who are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
* Has leptomeningeal carcinomatosis or metastasis
* Had prior treatment with:

  * Any agent including antibody drug conjugate (ADC) containing a chemotherapeutic agent targeting topoisomerase I
  * TROP2-targeted therapy
  * Docetaxel
* Had prior treatment with platinum-based chemotherapy and prior immunotherapy for Stage II NSCLC disease (eg, in the neo-adjuvant or adjuvant setting) without subsequently meeting the prior therapy requirements for Stage III or metastatic NSCLC disease
* Has NSCLC disease that is eligible for definitive local therapy alone
* Has uncontrolled or significant cardiac disease, including:

  * Mean QT interval corrected for heart rate using Fridericia's formula >470 msec (based on the average of Screening triplicate 12-lead electrocardiogram [ECG] determinations).
  * Myocardial infarction or uncontrolled/unstable angina within 6 months before randomization
  * Congestive heart failure (CHF) (New York Heart Association Class II to IV) at Screening. Participants with a history of Class II to IV CHF prior to Screening, must have returned to Class I CHF and have LVEF ≥50% (by either an ECHO or MUGA scan within 28 days before randomization) in order to be eligible.
  * Uncontrolled or significant cardiac arrhythmia
  * LVEF <50% by ECHO or MUGA scan within 28 days before randomization
  * Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) within 28 days before randomization
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months before randomization, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.), or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or prior pneumonectomy.
* Significant third-space fluid retention (for example ascites or pleural effusion) and is not amenable for required repeated drainage
* Clinically significant corneal disease
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals; suspected infections (eg, prodromal symptoms); or inability to rule out infections
* Has known human immunodeficiency virus (HIV) infection that is not well controlled
* Has an active or uncontrolled hepatitis B and/or hepatitis C infection, is positive for hepatitis B or C virus based on the evaluation of results of tests for hepatitis B (hepatitis B surface antigen [HBsAg], anti-hepatitis B surface antibody [anti-HBs], anti-hepatitis B core antibody [anti-HBc], or hepatitis B virus [HBV] DNA), and/or hepatitis C infection (as per hepatitis C virus [HCV] RNA) within 28 days of randomization.
* Has a history of malignancy, other than NSCLC, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥3 years
* Toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet improved to NCI-CTCAE version 5.0 Grade ≤1 or baseline
* Has a history of severe hypersensitivity reactions to either the drug substances, inactive ingredients (including but not limited to polysorbate 80) of DS-1062a or docetaxel, or monoclonal antibodies
* Pregnant or breastfeeding
* Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (209):
- United States (32):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - St. Joseph Heritage Healthcare, Anaheim, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - University of California San Diego, La Jolla, California
  - UCLA, Los Angeles, California
  - PIH Health, Whittier, California
  - Memorial Healthcare System- Memorial Cancer Institute, Hollywood, Florida
  - Orlando Health, Orlando, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ft. Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Baptist Health Louisville, Louisville, Kentucky
  - Baton Rouge General, Baton Rouge, Louisiana
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Meridian Hematology and Oncology, Manahawkin, New Jersey
  - Astera Cancer Care, Somerset, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Roger Williams Medical Center, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialist, Fairfax, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (4):
  - CER San Juan, Buenos Aires
  - Centro de Investigacion Pergamino S.A., Pergamino
  - Instituto de OncologÃƒÂ-a de Rosario, Rosario
  - Gaston Martinengo, Rosario
- Australia (6):
  - Flinders Medical Centre, Bedford Park
  - Blacktown Hosital, Blacktown
  - Austin Hospital, Heidelberg
  - Macquarie Hospital, North Ryde
  - Crown Princess Mary Cancer Centre Westmead Hospital, Sydney
  - Southern Medical Day Care Centre, Wollongong
- Belgium (4):
  - Centre Hospitalier Jolimont-Lobbes, Haine-Saint-Paul
  - CHA Centre Hospitalier de l Ardenne, Libramont
  - CHR site de la Citadelle, Liège
  - CHU UCL Namur, Yvoir
- Brazil (5):
  - Instituto do Cancer do Ceara - ICC, Fortaleza
  - Hospital Sao Lucas da Pucrs, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - Instituto Nacional de Cancer-INCA, Rio de Janeiro
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario
  - Sunnbrook Health Sciences Centre, Toronto, Ontario
  - MUHC-Glen Site and MUHC Research Institute, Montreal, Quebec
- China (19):
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital central south university, Changsha
  - Linyi Cancer Hospital, Hangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzou
  - Harbin Medical University Cancer Hospital, Heilongjiang
  - Jiamusi Cancer Tuberculosis Hospital, Heilongjiang
  - Fudan University Shanghai Cancer Center, Henan
  - Hubei Cancer Hospital, Hubei
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliated Hospital of Xi'an Jiaotong University, Shandong
  - Shanghai Chest Hospital, Shanghai
  - Henan Cancer Hospital, Shanghai Sheng
  - Zhejiang Cancer Hospital, Shanxi
  - West China Hospital, Sichuan University, Sichuan Province
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Zhejiang
- Vseobecna Fakultni Nemocnice VFN, Prague, Czechia
- France (13):
  - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Leon Berard, Lyon
  - CHU Louis Pradel, Lyon
  - APHM - Hopital Nord, Marseille
  - University Hospital of Nantes - Thoracic Oncology, Nantes
  - Institut Curie, Paris
  - CHU de Poitier Pole regional de Cancerologie, Poitiers
  - Hopital Pontchaillou, Rennes
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Hopital Foch, Sureesnes
  - CHU Toulouse Hopital Larrey, Toulouse
  - Gustav Roussy Cancer Campus Grand Paris, Villejuif
- Germany (11):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaet zu Koeln - Uniklinik Koeln, Cologne
  - IKF Krankenhaus Nordwest, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Fachklinik Muenchen-Gauting, Gauting
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Klinikverbund AllgÃ¤u, Kempten
  - Medizinische Klinik V, Standort Gießen
  - Klinikum Traunstein, Traunstein
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital / The Chinese University of Hong Kong, Hong Kong
- Hungary (5):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Szent Borbala Korhaz, Tatabánya
  - Tolna Megyei Balassa Janos Korhaz, Tolna
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (9):
  - Azienda Ospedaliero- Universitaria Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Policlinico G Rodolico San Marco, Catania
  - ASL 3 Genovese Oncologia Medica Villa Scassi, Genova
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Instituicao de Fisioterapeutas Ocupacionais, Roma
- Japan (21):
  - Hyogo Cancer Center, Akashi
  - Niigata Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Kansai Medical University Hospital, Hirakata
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Kyoto University Hospital, Kyoto
  - NHO Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-chō
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Saitama Cancer Center, Saitama
  - Sendai Kousei Hospital, Sendai
  - NHO Hokkaido Cancer Center, Shiroishi
  - Tokushima University Hospital, Tokushima
  - National Cancer Center Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
- Mexico (4):
  - San Peregrino Cancer Center, Aguascalientes
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Hospital Medica Sur Tlalpan, Mexico City
  - Hospital Universitario Jose Eleuterio Gonzalez, Monterrey
- Netherlands (4):
  - Erasmus MC, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Isala Klinieken, Harderwijk
  - St. Jansdal Ziekenhuis, Rotterdam
- Poland (9):
  - II Klinika Chorob Pluc i Gruzlicy, Bialystok
  - Szpitale Pomorskie Sp.zo.o, Gdynia
  - Ms Pneumed, Lublin
  - SP Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Med Polonia Sp. z o.o., Poznan
  - Szpital Specjalistyczny w Prabutach Sp. z o.o., Prabuty
  - Oddział Onkologii Wojewódzki Szpital Specjalistyczny Słupsk, Słupsk
  - Magodent Sp. z.o.o Szpital Elblaska, Warsaw
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- FDI Clinical Research, San Juan, Puerto Rico
- Romania (8):
  - SC Oncopremium Team SRL, Baia Mare
  - Institutul Oncologic Profesor Doctor Alexandru Trestioreanu, Bucharest
  - Centrul Medical Sanador, Bucharest
  - Clinical Emergency Hospital, Constanța
  - Onco Clinic Consult SA, Craiova
  - Sf Nectarie Oncology Center, Craiova
  - Oncolab SRL, Craiova
  - SC Oncomed SRL, Timișoara
- Russia (7):
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - Federal State Budgetary Institution - N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - University Headache Clinic LLC, Moscow
  - VitaMed LLC, Moscow
  - Institute of Oncology Hadassah Moscow, Moscow
  - LLC MSCH "Klinitsist", Novosibirsk
  - N.N. Petrov Research Institute of Oncology, Saint Petersburg
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - ICON Cancer Centre Farrer Park Hospital, Singapore
  - OncoCare Cancer Centre - Gleneagles Medical Centre Location, Singapore
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - St. Vincents Hospital The Catholic University of Korea, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
- Spain (13):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerte de Hierro de Majadahonda, Madrid
  - Hospital Regional Universitario Málaga, Málaga
  - CHUO, Ourense
  - Hospital Virgen Macarena, Seville
  - Hospital Universitario de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario Lozano Bleza, Zaragoza
- Switzerland (3):
  - Inselspital UniversitÃ¤tsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Waid ; Triemli, Site Triemli - clinic for Medical oncology & hematology, Zurich
- Taiwan (8):
  - E-Da Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital CGMH - Kaohsiung Branch, Niaosong
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital NCKUH, Tainan
  - Chi Mei Medical Center CMMC - Liouying Branch, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - LinKou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (3):
  - University College Hospital, London
  - The Christie Hospital, Manchester
  - The James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Sands J, Ahn MJ. Datopotamab deruxtecan versus docetaxel for non-small cell lung cancer: a plain language summary of the TROPION-Lung01 study. Future Oncol. 2025 Nov 21:1-14. doi: 10.1080/14796694.2025.2586004. Online ahead of print. PMID 41268710
- [Derived] Ahn MJ, Tanaka K, Paz-Ares L, Cornelissen R, Girard N, Pons-Tostivint E, Vicente Baz D, Sugawara S, Cobo M, Perol M, Mascaux C, Poddubskaya E, Kitazono S, Hayashi H, Hong MH, Felip E, Hall R, Juan-Vidal O, Brungs D, Lu S, Garassino M, Chargualaf M, Zhang Y, Howarth P, Uema D, Lisberg A, Sands J; TROPION-Lung01 Trial Investigators. Datopotamab Deruxtecan Versus Docetaxel for Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer: The Randomized, Open-Label Phase III TROPION-Lung01 Study. J Clin Oncol. 2025 Jan 20;43(3):260-272. doi: 10.1200/JCO-24-01544. Epub 2024 Sep 9. PMID 39250535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 605 participants , including 1 participant who was randomized twice, were randomized to the study in Europe, Asia, North America, South America, and Australia.
Groups:
- DS-1062a 6.0 mg/kg: Participants were randomized to receive 6.0 mg/kg of DS-1062a.
- Docetaxel 75 mg/m^2: Participants were randomized to receive 75 mg/m^2 docetaxel.
Period: Overall Study
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Started ("Started" signifies number of participants randomized) | 299 | 305
Completed ("Complete" signifies number of participants ongoing in study) | 68 | 62
Not Completed | 231 | 243
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 213 | 212
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 15 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2 | Total
Number analyzed (Participants) | 299 | 305 | 604
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 162 | 155 | 317
  >=65 years | 137 | 150 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.09) | 62.6 (10.28) | 62.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 95 | 211
  Male | 183 | 210 | 393
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 121 | 120 | 241
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 123 | 126 | 249
  Other | 42 | 47 | 89
  Unknown or Not Reported | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) As Assessed by Blinded Independent Central Review (BICR) Per RECIST v1.1 Following DS-1062a Versus Docetaxel
Description: PFS is defined as the time from randomization to the earlier of the dates of the first documentation of radiographic progressive disease or death due to any cause.
Time Frame: From randomization until disease progression or death (whichever occurs first), up to approximately 27 months
Population: Full Analysis Set includes all randomized subjects. If a subject was randomized more than once, only one of the participants is included in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 299 | 305
months | 4.4 [4.2 to 5.6] | 3.7 [2.9 to 4.2]

2. Primary Outcome: Overall Survival (OS) Following DS-1062a Versus Docetaxel
Description: OS is defined as the time from randomization to the date of death due to any cause.
Time Frame: From randomization until date of death due to any cause, up to to approximately 38 months
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: months
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 299 | 305
months | 12.9 (11.0) | 11.8 (10.1)

3. Secondary Outcome: Progression-free Survival (PFS) As Assessed by Investigator Per RECIST v1.1 Following DS-1062a Versus Docetaxel
Description: as for outcome 1
Time Frame: From randomization until disease progression or death (whichever occurs first), up to approximately 43 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 299 | 305
months | 4.4 [4.2 to 5.5] | 3.0 [2.8 to 4.0]

4. Secondary Outcome: Objective Response Rate (ORR) As Assessed by Blinded Independent Central Review (BICR) and Investigator As Per RECIST v1.1 Following DS-1062a Versus Docetaxel
Description: ORR is defined as the proportion of subjects who achieved a best overall response (BOR) of complete response (CR) or partial response (PR), as assessed by BICR and investigator per RECIST v1.1.
Time Frame: From randomization until disease progression or death (whichever occurs first), up to approximately 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 299 | 305
Participants
  Assessed by Blinded Independent Central Review | 79 | 39
  Assessed by Investigator | 74 | 44

5. Secondary Outcome: Duration of Response (DOR) As Assessed by Blinded Independent Central Review (BICR) and Investigator As Per RECIST v1.1 Following DS-1062a Versus Docetaxel
Description: DOR is defined as the time from the date of the first documentation of objective response (confirmed CR or confirmed PR) to the date of the first documentation of radiographic Progressive Disease or death due to any cause, whichever occurs first.
Time Frame: From date of first objective response (CR or PR) to date of first radiographic disease progression or death due to any cause (whichever occurs first), up to approximately 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 299 | 305
months
  Assessed by Blinded Independent Central Review | 7.1 [5.6 to 10.9] | 5.6 [5.4 to 8.1]
  Assessed by Investigator | 9.6 [6.7 to 11.1] | 6.4 [5.1 to 8.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 28 days after last dose of the study drug, up 43 months.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE with a start or worsening date on or after the start date of study treatment until 35 days since date of last dose of study treatment. Adverse Events used Safety Analysis Set, while Mortality used Full Analysis Set.
Arm/Group | DS-1062a 6.0 mg/kg | Docetaxel 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 215/299 | 218/305
Serious Adverse Events (participants affected / at risk) | 92/297 | 111/290
Other Adverse Events (participants affected / at risk) | 273/297 | 262/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DS-1062a 6.0 mg/kg (N=297) | Docetaxel 75 mg/m^2 (N=290)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 11 (11)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (3) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 3 (5)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 5 (6) | 8 (9)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0/0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pericarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 15 (19) | 23 (26)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia serratia (Infections and infestations) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intrac (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0/0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 6 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DS-1062a 6.0 mg/kg (N=297) | Docetaxel 75 mg/m^2 (N=290)
Anaemia (Blood and lymphatic system disorders) | 50 (90) | 72 (140)
Leukopenia (Blood and lymphatic system disorders) | 6 (7) | 20 (32)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 40 (66)
Dry eye (Eye disorders) | 21 (23) | 3 (3)
Lacrimation increased (Eye disorders) | 23 (23) | 17 (17)
Constipation (Gastrointestinal disorders) | 58 (70) | 42 (47)
Diarrhoea (Gastrointestinal disorders) | 38 (54) | 65 (90)
Dry mouth (Gastrointestinal disorders) | 16 (20) | 9 (9)
Nausea (Gastrointestinal disorders) | 112 (166) | 54 (74)
Stomatitis (Gastrointestinal disorders) | 148 (279) | 47 (65)
Vomiting (Gastrointestinal disorders) | 47 (65) | 26 (37)
Asthenia (General disorders) | 70 (139) | 69 (107)
Chest pain (General disorders) | 17 (19) | 12 (12)
Fatigue (General disorders) | 48 (59) | 48 (70)
Malaise (General disorders) | 21 (34) | 30 (45)
Oedema peripheral (General disorders) | 13 (15) | 40 (56)
Pyrexia (General disorders) | 22 (25) | 35 (49)
COVID-19 (Infections and infestations) | 34 (38) | 23 (23)
Conjunctivitis (Infections and infestations) | 15 (19) | 3 (3)
Pneumonia (Infections and infestations) | 20 (25) | 12 (13)
Alanine aminotransferase increased (Investigations) | 16 (30) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 15 (27) | 8 (14)
Blood creatinine increased (Investigations) | 16 (21) | 4 (5)
Neutrophil count decreased (Investigations) | 9 (27) | 41 (99)
Weight decreased (Investigations) | 28 (37) | 13 (16)
White blood cell count decreased (Investigations) | 6 (15) | 27 (60)
Decreased appetite (Metabolism and nutrition disorders) | 86 (119) | 63 (70)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (25) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (36) | 33 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (23) | 17 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 25 (33)
Dysgeusia (Nervous system disorders) | 17 (18) | 14 (17)
Headache (Nervous system disorders) | 28 (35) | 14 (15)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 28 (45)
Paraesthesia (Nervous system disorders) | 4 (4) | 18 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 15 (19)
Insomnia (Psychiatric disorders) | 15 (16) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (56) | 37 (46)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 (65) | 46 (55)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 15 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 95 (115) | 101 (115)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (21) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (40) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 40 (45) | 21 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT04656652/Prot_SAP_000.pdf